CLINICAL TRIAL: NCT04508738
Title: Effects of Combined Interventions to Optimize Recovery During High-intensity Exercises in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ERP_2020
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2020-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Each participant will be tested on 4 different days with a control, a placebo and an interventional condition in random order.
Who Masked: Participant
Masking Description: Participants will be blinded about the true nature of the placebo intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ERP Intervention (Experimental): Combination of different methods to improve recovery.
  Interventions: Other: ERP
- Control (No Intervention): Passive recovery by sitting on a chair
- Placebo (Placebo Comparator): A combination of methods similar to the ERP intervention but at an intensity / mixture supposed to be ineffective at improving recovery.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: ERP — The ERP intervention is applied in a randomized and counter-balanced order across visits 2-4 in each 3-min break in-between the six 30-s sprints, with one intervention per visit. The order and timing of the constituents of the interventions will be strictly constant within and between participants.
  ERP: 1) neck cooling with an iced gel pad, 2) drinking a ∼ 6% CHO solution, 3) mouth-rinsing with a ∼10% CHO, ∼6 mg ･ kg -1 caffeine solution, 4) performing submaximal squats and 5) hyperventilating a hyperoxic mixture
  Arms: ERP Intervention
Other: Placebo — The control intervention is applied in a randomized and counter-balanced order across visits 2-4 in each 3-min break in-between the six 30-s sprints, with one intervention per visit. The order and timing of the constituents of the interventions will be strictly constant within and between participants.
  1) neck "cooling" with room temperature gel pack, 2) drinking an artificially sweetened solution, 3) mouth-rinsing with artificially sweetened solution (containing no caffeine), 4) performing unloaded squat manoeuvres, 5) deep breaths with room air
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the effects a complex recovery intervention during the breaks of a repeated sprint test on exercise performance compared to placebo and control conditions. The enhanced recovery package (ERP) includes neck cooling with an iced gel pad, drinking a 6% CHO solution, mouth-rinsing with a 10% CHO, 6 mg･kg -1 caffeine solution, performing submaximal squats and hyperventilating a hyperoxic mixture; all applied in each 3-min break in-between the six 30-s sprints. This intervention will be compared to a placebo and a control condition.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Healthy
* Male
* Age: 18-40 years
* Body-Mass-Index (BMI): 18.5-24.9 kg･m-2
* Trained individuals: max. Power output ≥ 4.0 Watts･kg-1
* Non-smoking
* Willingness to adhere to the study rules

Exclusion Criteria:

* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participants
* Previous enrolment into the current study
* Intake of medications affecting performance or the respiratory, cardiovascular or neuromuscular system
* Acute or chronic illness affecting performance or the respiratory, cardiovascular or neuromuscular system

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in mean power output | through study completion, an expected average of 3 weeks per participant
  Measured over the six 30s high-intensity cycling sprints in each of the three conditions. Mean power mirrors the body's ability to generate muscle power and physical energy. Any meaningful effects of the recovery interventions will eventually translate into a higher power output.
Change in fatigue index | through study completion, an expected average of 3 weeks per participant
  Fatigue index = drop in power output from the beginning to the end a 30s sprint test. The change in this index will be calculated from the 1st to the 6th sprint test in each condition.

CONTACTS AND LOCATIONS:
Overall Officials: Christina M. Spengler, Prof., Principal Investigator — Christina M. Spengler, Prof. Study Principal Investigator Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich
Locations (1):
- ETH Zürich, Exercise Physiology Lab, Zurich, Canton of Zurich, Switzerland